CLINICAL TRIAL: NCT05006469
Title: Observation of the Efficacy of BAd Regimen in the Treatment of Relapsed and Refractory Multiple Myeloma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Liao Aijun (Other)
Responsible Party: Sponsor-Investigator, Liao Aijun, Director of Hematology, Shengjing Hospital
Organization: Shengjing Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021PS168J
Record Dates: First submitted 2021-08-02; First posted 2021-08-16 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-08

CONDITIONS: Bendamustine; Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Bendamustine Hydrochloride; Doxorubicin; Dexamethasone

STUDY DESIGN:
Intervention Model Description: Relapsed and refractory MM received bendamustine combined with liposomal adriamycin (or adriamycin) and dexamethasone (BAd) for treatment
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BAd treatment (Experimental): Bendamustine 70-90mg/m2, d1, d2 Liposome Adriamycin 15-20mg/m2, d1 or Adriamycin 10mg d1-d4 Dexamethasone 40mg qw po. (20mg, >70 years old) There is a course of treatment every 28 days, and a total of 6 courses are completed.
  Interventions: Drug: Bendamustine

INTERVENTIONS:
Drug: Bendamustine — Bendamustine 70-90mg/m2, d1, d2 Liposome Adriamycin 15-20mg/m2, d1 or Adriamycin 10mg d1-d4 Dexamethasone 40mg qw po. (20mg, >70 years old) There is a course of treatment every 28 days, and a total of 6 courses are completed.
  Other Names: Liposome Adriamycin; Adriamycin; dexamethasone

SUMMARY:
Observe the best dose, efficacy and adverse reactions of BAd in the treatment of relapsed and refractory multiple myeloma.

DETAILED DESCRIPTION:
Multiple myeloma (MM) is the second most common malignant tumor of the hematological system, accounting for 10% of all hematological malignancies. With the emergence of new drugs such as proteasome inhibitors and immunomodulators, the efficacy of MM has been significantly improved, and the progression-free survival rate and overall survival rate of patients have been significantly improved. However, due to primary or secondary drug resistance, MM is still incurable , and patients will eventually be relapsed and refractory. At present, most first-line treatments contain proteasome inhibitors and immunomodulators at the same time, and patients are often resistant to these two types of drugs. CD38 monoclonal antibody is a new drug that was launched two years ago, but the price is too high, roughly 500,000 yuan a year, and most patients cannot afford it. At present, new drugs available to patients in China is still very limited, and investigator urgently need to find new treatment options among the existing drugs in China to prolong the lives of patients. Bendamustine is an alkylating agent and is currently mainly used in the treatment of lymphoma in China. But in Europe, bendamustine has been approved as a MM drug. The NCCN guidelines also include bendamustine + proteasome inhibitors or immunomodulators + hormones as the recommended treatment for MM. Because most of the patients with relapse and refractory MM have been resistant to proteasome inhibitors and immunomodulators, investigator found that the NCCN guidelines recommended schemes are not effective when used in these patients. Therefore, investigator tried to combine bendamustine with liposomes and dexamethasone (BAd) to treat relapsed and refractory MM. At present, 3 patients have been treated with this program, all of which are multi-line recurrences. Among them, 1 patient achieved complete response (CR) after 2 courses of treatment. At present, 6 courses of treatment have been completed and have been in CR state. The other 2 cases achieved partial response, and the total response rate reached 100%. The common adverse reaction in patients was hematological toxicity, but they were all tolerated. No patient stopped the drug due to adverse reactions. The price of bendamustine per course of treatment is roughly between 6000-8000 yuan, which patients can basically afford. Therefore, the program is feasible in terms of effectiveness, economy and safety. Due to the small number of patients, investigator need to further expand the number of samples to observe the optimal dose, efficacy and adverse reactions of the drug. If the program is validated and feasible, it will benefit more patients, extend their lives as much as possible, and have the opportunity to wait for other new drugs to come out.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old
2. ≥1 line relapsed or refractory multiple myeloma
3. Alanine aminotransferase is less than 2.5 times the upper limit of normal, and total bilirubin is less than 1.5 times the upper limit of normal
4. Creatinine clearance rate>40ml/min
5. No serious heart disease

Exclusion Criteria:

1. Untreated multiple myeloma patients
2. Pregnant or lactating women
3. Alanine aminotransferase is more than 2.5 times the upper limit of normal, and total bilirubin is more than 1.5 times the upper limit of normal
4. Creatinine clearance rate ≤40ml/min
5. Severe heart disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-05-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
ORR, CR, PR, MR, SD | From the start of the treatment to the end of the 6-course treatment
  Overall response rate (ORR), complete response (CR) ,partial response (PR) ,micro response (MR) and stable disease（SD）are calculated to evaluate the efficacy;
The rate of adverse event | From the start of the treatment to the end of the 6-course treatment
  Safety was evaluated based on hematology, nonhematology adverse events,such as thrombocytopenia,nausea,vomit.

SECONDARY OUTCOMES:
survival | From the start of the treatment until the disease progresses.If the patient has no disease progression, the follow-up time will end 1 year after the treatment
  Progress free survival (PFS) is calculated to evaluate survival status.

CONTACTS AND LOCATIONS:
Overall Officials: Liao Aijun, Study Director — Shengjing Hospital
Locations (1):
- Shengjing Hospital of China Medical University, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No